CLINICAL TRIAL: NCT03045289
Title: Whole-Food, Plant-Based Nutrition Among Women With Metastatic Breast Cancer: A Pilot Study of Recruitment, Retention, and Preliminary Changes in Biomarkers and Symptoms.
Brief Title: A Whole-food, Plant-Based Nutrition Intervention in Women With Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Thomas M Campbell, Instructor of Clinical Family Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSRB00066846
Record Dates: First submitted 2017-02-01; First posted 2017-02-07 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Breast Cancer; Breast Cancer Stage IV
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet, Plant-Based

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Subjects are provided three meals daily, attend weekly office visits, take a daily multivitamin.
  Interventions: Behavioral: Plant-Based Diet
- Control Group (No Intervention): Women instructed to maintain current intake and take a provided multivitamin.

INTERVENTIONS:
Behavioral: Plant-Based Diet — Women will be provided with 3 meals daily, delivered to their home, for 8 weeks, along with a multivitamin, and will attend weekly office visits.
  Arms: Intervention group

SUMMARY:
This research will examine the feasibility of conducting a strict whole-food, plant-based dietary intervention in women with stable metastatic breast cancer currently undergoing conventional treatments. In addition, this research will provide preliminary data on dietary intakes and the effect of plant-based nutrition on numerous outcomes reflecting cancer prognosis and overall health using advanced imaging, various blood biomarkers linked to cancer progression, and numerous symptom questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women with a confirmed diagnosis of metastatic breast cancer with a stable treatment regimen, demonstrated by no changes in primary cancer therapy 6 weeks prior to consent and no anticipated changes in primary cancer therapy in the 4 weeks following consent.
* Systemic therapy may consist of any conventional treatment including anti-hormonal, cytotoxic, targeted monoclonal antibody or small molecule kinase inhibitors or any combination of the above. Women who have previously declined conventional cancer therapy are also eligible provided they meet all other eligibility criteria.
* Expected to survive for at least 6 months.
* Eligibility classification for enrollment into the study - T: any; N: any; M:1.
* Any ER/PR/HER2 status is eligible.
* Age > 18 years.
* Must be willing to adopt a strict, whole-foods, plant-based diet.
* Participant must be willing and able to comply with the protocol for the duration of the study including scheduled testing and weekly office visits.
* Able to speak and read English fluently.

Exclusion Criteria:

* Inability to tolerate a normal diet.
* Current use of insulin or sulfonylureas.
* Active malabsorption syndrome at time of consent (ie. Crohn's disease, major bowel resection leading to permanent malabsorption).
* Current eating disorder.
* Uncontrolled diarrhea.
* Plant-based food allergies or intolerances.
* Recent consumption (in the past 6 months) of a vegan diet.
* GFR < 30 on 2 or more lab tests in the past 90 days.
* Serum potassium > 5.3 on 2 or more lab tests in the past 90 days.
* Major surgery within 2 months of starting study program.
* Psychiatric disorder that prohibits giving informed consent.
* Current smoking.
* Current high risk alcohol use (> 7 drinks per week).
* Current illicit substance use.
* Current warfarin use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women will be enrolled due to low numbers of male breast cancer patients and inability to create subgroup analyses.
Enrollment: 32 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Recruitment | 1 year
  Percentage of women who are randomized in the study out of the all women approached.
Retention | 8 weeks
  Percentage of women who start the intervention who go on to complete 8-week testing
Compliance | 8 weeks
  The percentage of daily calorie intake from "on-plan" food will be calculated for each participant.

SECONDARY OUTCOMES:
FACT-B | 8 weeks
EORTC QLQ-C30 | 8 weeks
FACT-COG | 8 weeks
Brief Fatigue Inventory (BFI) | 8 weeks
Symptom Inventory | 8 weeks
Serum breast cancer biomarkers | 8 weeks
  CA 15-3, CEA, CA 27.29
Tumor Metabolic Activity as assessed by Positron Emission Tomography/ Computer Tomography (PET/CT) | 8 weeks
Changes in nutrient intakes based on 3 day food diaries | 8 weeks
  Assess baseline diet compared to intervention diet
Weight | 8 weeks
Blood Pressure | 8 weeks
Inflammatory Markers | 8 weeks
  CBC, CRP
Hormonal Levels | 8 weeks
  Estradiol, testosterone, SHBG, DHEAS, Insulin, IGF-1, IGFBP-3
Metabolic Markers | 8 weeks
  Lipids, CMP
Tumor Metabolic Activity | 8 weeks
  PET/CT scan SUV Uptake
Circulating Tumor Cells | 8 weeks
cell-free DNA | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Campbell, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be made available for collaboration or other purposes with appropriate data use agreements in place.

REFERENCES:
- [Derived] Scales TQ, Smith B, Blanchard LM, Wixom N, Tuttle ET, Altman BJ, Peppone LJ, Munger J, Campbell TM, Campbell EK, Harris IS. A whole food, plant-based diet reduces amino acid levels in patients with metastatic breast cancer. Cancer Metab. 2024 Dec 19;12(1):38. doi: 10.1186/s40170-024-00368-w. PMID 39702320
- [Derived] Scales TQ, Smith B, Blanchard LM, Wixom N, Tuttle ET, Altman BJ, Peppone LJ, Munger J, Campbell TM, Campbell EK, Harris IS. A whole food, plant-based diet reduces amino acid levels in patients with metastatic breast cancer. medRxiv [Preprint]. 2024 Oct 22:2024.10.09.24315165. doi: 10.1101/2024.10.09.24315165. PMID 39417128
- [Derived] Campbell EK, Campbell TM, Culakova E, Blanchard L, Wixom N, Guido JJ, Fetten J, Huston A, Shayne M, Janelsins MC, Mustian KM, Moore RG, Peppone LJ. A whole food, plant-based randomized controlled trial in metastatic breast cancer: feasibility, nutrient, and patient-reported outcomes. Breast Cancer Res Treat. 2024 Jul;206(2):273-283. doi: 10.1007/s10549-024-07284-z. Epub 2024 Mar 30. PMID 38553649
- [Derived] Campbell TM, Campbell EK, Culakova E, Blanchard LM, Wixom N, Guido JJ, Fetten J, Huston A, Shayne M, Janelsins MC, Mustian KM, Moore RG, Peppone LJ. A whole-food, plant-based randomized controlled trial in metastatic breast cancer: weight, cardiometabolic, and hormonal outcomes. Breast Cancer Res Treat. 2024 Jun;205(2):257-266. doi: 10.1007/s10549-024-07266-1. Epub 2024 Mar 6. PMID 38446316
- [Derived] Campbell EK, Campbell TM, Culakova E, Blanchard LM, Wixom N, Guido J, Fetten J, Huston A, Shayne M, Janelsins M, Mustian K, Moore RG, Peppone LJ. A Whole Food, Plant-Based Randomized Controlled Trial in Metastatic Breast Cancer: Feasibility, Nutrient, and Patient-Reported Outcomes. Res Sq [Preprint]. 2023 Nov 21:rs.3.rs-3606685. doi: 10.21203/rs.3.rs-3606685/v1. PMID 38045318
- [Derived] Campbell TM, Campbell EK, Culakova E, Blanchard L, Wixom N, Guido J, Fetten J, Huston A, Shayne M, Janelsins MC, Mustian KM, Moore RG, Peppone LJ. A Whole-Food, Plant-Based Randomized Controlled Trial in Metastatic Breast Cancer: Weight, Cardiometabolic, and Hormonal Outcome. Res Sq [Preprint]. 2023 Nov 8:rs.3.rs-3425125. doi: 10.21203/rs.3.rs-3425125/v1. PMID 37986940